CLINICAL TRIAL: NCT04093960
Title: A Randomized, Double-blind, Comparison of the Efficacy and Safety of Escitalopram Plus PS128 to Escitalopram in the Acute Treatment of Patients With Major Depressive Disorder
Brief Title: Escitalopram Plus PS128 vs. Escitalopram
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Ching-Hua Lin, MD, PhD, Chief of Adult Psychiatry, Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSPH-2016-02
Record Dates: First submitted 2019-09-02; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Major Depression
Keywords: psychobiotics; major depressive disorder; escitalopram
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- escitalopram plus128 (Experimental): escitalopram (10 mg daily) plus PS128(a psychobiotic) (300 mg two times daily, equivalent to 3 ×1010 CFU two times daily)
  Interventions: Dietary Supplement: Lactobacillus plantarum PS128
- escitalopram (Active Comparator): 10 mg/d of escitalopram
  Interventions: Dietary Supplement: Lactobacillus plantarum PS128

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum PS128 — 10 mg qd of escitalopram qd plus 300mg bid of Lactobacillus plantarum PS128 to enhance antidepressive effect

SUMMARY:
The purpose of this study is to compare the efficacy and safety of escitalopram plus PS128 to escitalopram in the acute treatment of patients with major depressive disorder.

DETAILED DESCRIPTION:
In this 6-week, double-blind, fixed-dose study, patients with major depressive disorder are randomly assigned to escitalopram (10 mg daily) plus PS128 (a psychobiotic) (300 mg two times daily, equivalent to 3 ×1010 CFU two times daily) or escitalopram (10 mg daily) groups. The rating scales and instrument, including Clinical Global Impression-Severity, 17-item Hamilton Rating Scale for Depression, Hamilton Anxiety Rating Scale, Global Assessment of Functioning, Heart Rate Variability, Depression and Somatic Symptoms Scale, Work and Social Adjustment Scale, Short form 36 and Pittsburgh Sleep Quality Index, are used to measure treatment outcomes at weeks 0, 1, 2, 3, 4, 5, and 6. UKU Side Effect Rating Scale and Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome are used to measure side effects. Generalized estimating equations model will be used to analyze the differences between two groups with respect to efficacy and safety measures on time after adjusting for baseline severity, sex, age and age at onset of illness.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder
* CGI >=4
* the score of the 17-item Hamilton Rating Scale for Depression (HAMD-17) was 18 or higher.
* washout of antipsychotics at least 3 days
* written informed consents
* Not taking fluoxetine at least one month before admission.

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder or organic mental disorders.
* comorbid with substance abuse/dependence in the past 6 months.
* with psychotic features
* treatment-resistant depression or receiving electroconvulsive therapy.
* History of serious adverse events to escitalopram
* female subjects with pregnancy or lactation.
* severe physical illness
* receiving antibiotics treatment in the past two weeks.
* taking products with probiotics.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Depression severity by the change of 17-item Hamilton Rating Scale for Depression (HAMD-17) total scores | Time Frame: The HAMD-17 was rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  17-item Hamilton Rating Scale for Depression (HAMD-17) is widely used in clinical setting to evaluate depression symptoms in the past week. Higher total HAMD-17 scores (ranging from 0 to 52) indicate more severe depression.

SECONDARY OUTCOMES:
Clinical severity by Clinical Global Impression-Severity (CGI-S) | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  The CGI was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI comprises one-item measures evaluating the severity of psychopathology from 1 to 7 and higher scores indicate higher severity.
Assessments of safety for general adverse events | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  General adverse events were evaluated by a standardized the UKU Side Effect Rating Scale. A score of 1, 2 or 3 on any UKU item that first occurred or worsened during treatment indicated adverse events "cases".
Change of body weights | Time Frame: Body weights were assessed at baseline and week 6(or on early termination).
  Body weights
Change of body mass index (BMI) | Time Frame: BMI was assessed at baseline and week 6(or on early termination).
  body mass index (BMI)
Change of pulse rate | Time Frame: Pulse rates were checked at baseline and at weeks 1, 2, 3, 4, and 6 (or on early termination).
  pulse rate
Change of blood pressure | Time Frame: Blood pressure were checked at baseline and at weeks 1, 2, 3, 4, and 6 (or on early termination).
  blood pressure (both systolic and diastolic)
Change of ECG QT Interval | Time Frame: ECG were assessed at baseline and week 6 (or on early termination).
  12-lead electrocardiogram (ECG) ECG QT Interval.
change of fasting glucose. | Time Frame: laboratory test mentioned above were assessed at baseline and week 6(or on early termination.
  Laboratory tests including fasting glucose.
change of liver function | Time Frame: laboratory test mentioned above were assessed at baseline and week 6 (or on early termination).
  Laboratory tests including alanine aminotransferase [ALT] and aspartate aminotransferase [AST].
change of renal function | Time Frame: laboratory test mentioned above were assessed at baseline and week 6 (or on early termination).
  Laboratory tests including blood urea nitrogen [BUN], creatinine.
change of lipid profiles. | Time Frame: laboratory test mentioned above were assessed at baseline and week 6(or on early termination).
  Laboratory tests including triglycerides, cholesterol, high density lipoprotein [HDL], and low density lipoprotein [LDL].
Assessments of quality of life | Time Frame: Medical Outcomes Study Short-Form 36 was assessed at baseline and week 6
  The Short-Form-36 (SF-36) is comprised of the physical component summary (PCS) which measures physical health, and the mental component summary (MCS) which measures mental health. PCS includes 4 subscales: 1) physical functioning, 2) role physical limitations, 3) body pain, 4) general health; MCS includes 4 subscales: 1) vitality, 2) social functioning, 3) role emotional limitations, and 4) mental health. SF-36 raw scores were processed according to the user manual to obtain standardized scores for all 8 SF-36 subscales, PCS and MCS. Scores for the SF-36 subscales range from 0 to 100, with a higher score representing better QOL. The PCS and MCS were standardized according to general population means and variances to produce scores with a common mean of 50 and standard deviation of 10 (T-scores). Thus, any score < 50 represents a reduction from "normal" health.
Assessments of heart rate variability | Time Frame: Heart rate variability was assessed at baseline and week 6
  Heart rate variability
depression and somatic symptoms evaluation | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  The Depression and Somatic Symptoms Scale (DSSS) is composed of a 12-item depression subscale (DS) and a ten-item somatic subscale (SS), which includes a five-item pain subscale (PS). Each item is scored from 0 to 3 (absent, mild, moderate, and severe) according to the severity of symptoms, with the total score ranging from 0 to 36 and 0-30 for the DS and the SS, respectively. Higher total score indicates more severe depression and somatic symptoms.
Gastrointestinal Symptoms evaluation | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome (GSRS) includes 15 questions on a scale of 1 to 7, depending on how inconvenient it had been during the previous week. A higher score indicates more inconvenient symptoms. Combination scores among 15 questions can assess the following five domains: reflux syndrome (heartburn and acid regurgitation), abdominal pain (stomach ache, gastric hunger pains and nausea), indigestion syndrome (gastric borborygmus, gastric bloating, eructation and increased flatus), diarrhea syndrome (diarrhea, loose stools and urgent need to defecate) and constipation syndrome (constipation, hard stools and feeling of incomplete evacuation).
Sleep Quality evaluation: The Pittsburgh Sleep Quality Index (PSQI) | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The 19 items are grouped into 7 components, including (1) sleep duration, (2) sleep disturbance, (3) sleep latency, (4) daytime dysfunction due to sleepiness, (5) sleep efficiency, (6) overall sleep quality, and (7) sleep medication use. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality. In distinguishing good and poor sleepers, a global PSQI score > 5 yields a sensitivity of 89.6% and a specificity of 86.5%.
Function evaluation | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  Global Assessment of Functioning (GAF) is used to rate severity of illness in psychiatry and covers the range from positive mental health to severe psychopathology. It is an overall (global) measure of how patients are doing Internationally, recording GAF is either done with a single value (this is the most severe of the symptom and functioning values) or both symptom (GAF-S) and functioning (GAF-F) values are recorded. The symptom and functioning scales have both 100 scoring possibilities (1-100). The 100-point scales are divided into 10 intervals, or sections, each with 10 scoring possibilities (examples: 31-40 and 51- 60). Verbal instructions (called anchor points) describe symptoms and functioning relevant for scoring in the 10-point intervals.
change of work and social adjustment | The scales were rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination).
  Work and Social Adjustment Scale(WSAS) is a widely used questionnaire by patients' perspectives concerning impaired functioning. The WSAS comprises 5 items (work, home management, social leisure, private leisure, and relationships; see Appendix A), each rated on a scale of 0 to 8, which can also be pooled (total score 0-40; higher scores denote more disability)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Municipal Kai-Syuan Psychiatric Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided